CLINICAL TRIAL: NCT07242404
Title: Evaluation of Agreement Between the Handheld Elastography Device and iLivTouch for Multi-Position Liver Assessment in Chronic Liver Disease
Brief Title: Comparison of a Handheld Elastography Device With iLivTouch in Chronic Liver Disease Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Hong You (Other)
Responsible Party: Sponsor-Investigator, Hong You, Principal Investigator, Beijing Friendship Hospital
Organization: Beijing Friendship Hospital (Other)
Other Study IDs: 2025-P2-511-01
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: MAFLD; HEPATITIS B CHRONIC
Keywords: Transient Elastography; Noninvasive Liver Assessment; Agreement Study
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic Liver Disease Cohort: Adults with chronic hepatitis B and/or MASH receiving paired liver elastography assessments for agreement analysis.

SUMMARY:
This single-center cross-sectional study aims to evaluate the agreement between a handheld elastography device and the iLivTouch transient elastography system for the noninvasive assessment of liver fibrosis and steatosis in adults with chronic liver disease. The study compares liver stiffness measurement (LSM) and ultrasound attenuation parameter (UAP) obtained by both devices in the standard supine position, and further explores the feasibility and consistency of measurements performed in the sitting position.

All participants will undergo paired examinations using both devices in two body positions (supine and sitting). Agreement between devices and between body positions will be assessed using Bland-Altman analysis, intraclass correlation coefficients, and categorical consistency metrics. The study will also evaluate device performance indicators, including measurement success rate, procedure time, and battery endurance under simulated clinical conditions.

This study aims to provide clinical evidence on the accuracy, reliability, and feasibility of a new handheld transient elastography device, and to explore whether sitting-position measurements can serve as an alternative to standard supine assessment in chronic liver disease patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.
* Diagnosed with one of the following:

  * Chronic hepatitis B or compensated HBV-related cirrhosis (based on the 2022 Chinese CHB guidelines), or
  * Metabolic dysfunction-associated fatty liver disease (MAFLD), metabolic dysfunction-associated steatohepatitis (MASH), or fibrosis/cirrhosis due to MAFLD (based on the 2024 MAFLD guidelines).
* Willing and able to provide written informed consent.

Exclusion Criteria:

* Chronic liver disease due to other etiologies (e.g., other viral hepatitis, autoimmune liver disease, alcoholic liver disease, genetic/metabolic liver disease).
* Evidence of decompensated cirrhosis.
* Total bilirubin > 51 μmol/L.
* ALT > 5 × upper normal limit.
* Presence of hepatocellular carcinoma, hepatic hemangioma, large hepatic cyst, or other space-occupying liver lesions.
* Co-infection with HIV.
* History of liver transplantation or TIPS.
* Pregnancy.
* Congestive hepatopathy.
* Unhealed wounds in the right upper abdomen.
* Inability to maintain the required sitting position.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with chronic liver disease, including chronic hepatitis B, compensated HBV-related cirrhosis, and metabolic dysfunction-associated fatty liver disease (MAFLD), who undergo paired liver elastography measurements using two devices.
Sampling Method: Non-Probability Sample
Enrollment: 224 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Agreement Between the Handheld Elastography Device and iLivTouch for Liver LSM in the Supine Position | At the time of liver elastography assessment (baseline)

SECONDARY OUTCOMES:
ICC for LSM and UAP in the Supine Position | At baseline
Categorical Agreement in Fibrosis Staging and Steatosis Grading | At baseline
Agreement Between Devices in the Sitting Position | At baseline
Agreement Between Supine and Sitting Measurements (Handheld Device) | At baseline